CLINICAL TRIAL: NCT07155980
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled Ascending Dose Study to Evaluate the Safety, Tolerability and Pharmacology of GSM-779690T in Healthy Adult Participants
Brief Title: A Clinical Trial to Study Single- and Multiple- Doses of GSM-779690T in Healthy Participants
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: The protocol is being withdrawn prior to enrollment due to a redesign of the study approach under the existing IND.
Sponsor: Acta Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: ACT-C501
Record Dates: First submitted 2025-08-13; First posted 2025-09-04 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Healthy Adult Participants
Keywords: gamma-secretase modulator; Alzheimer's disease; Pharmacokinetics; pharmacodynamics; beta-amyloid; single ascending dose; multiple ascending dose
MeSH Terms: conditions — Plaque, Amyloid

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The active drug and placebo control have the same appearance and weight. The study drug or placebo will be prepared by a licensed pharmacist and dispense the active or placebo capsules to the participants according to the randomization schedule.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (10):
- Cohort 01: 20 mg (Experimental): Healthy adult participants receiving a single dose in the SAD study.
  Interventions: Drug: GSM-779690T; Other: Placebo
- Cohort 02: dose to be determined (Experimental): Healthy adult participants receiving a single dose in the SAD study.
  Interventions: Drug: GSM-779690T; Other: Placebo
- Cohort 03: dose to be determined (Experimental): Healthy adult participants receiving a single dose in the SAD study.
  Interventions: Drug: GSM-779690T; Other: Placebo
- Cohort 04: dose to be determined (Experimental): Healthy adult participants receiving a single dose (x2) in the SAD study.
  Interventions: Drug: GSM-779690T; Other: Placebo
- Cohort 05: dose to be determined (Experimental): Healthy adult participants receiving a single dose (x2) in the SAD study.
  Interventions: Drug: GSM-779690T; Other: Placebo
- Cohort 06: dose to be determined (Experimental): Healthy adult participants receiving a single dose in the SAD study.
  Interventions: Drug: GSM-779690T; Other: Placebo
- Cohort 07: dose TBD (Experimental): Healthy adult participants receiving a multiple dose in the MAD study.
  Interventions: Drug: GSM-779690T; Other: Placebo
- Cohort 08: dose TBD (Experimental): Healthy adult participants receiving a multiple dose in the MAD study.
  Interventions: Drug: GSM-779690T; Other: Placebo
- Cohort 09: dose TBD (Experimental): Healthy adult participants receiving a multiple dose in the MAD study.
  Interventions: Drug: GSM-779690T; Other: Placebo
- Cohort 10: dose TBD (Experimental): Healthy older-adult participants receiving a multiple dose in the MAD study.
  Interventions: Drug: GSM-779690T; Other: Placebo

INTERVENTIONS:
Drug: GSM-779690T — Opaque capsules for oral consumption.
Other: Placebo — Opaque capsules for oral consumption.

SUMMARY:
This is a randomized, double-blinded, placebo-controlled dose escalating first in human study to evaluate the safety, tolerability, pharmacokinetic (PK), pharmacodynamic (PD) of GSM-779690T. The study will have two parts: a single ascending dose (SAD) component and a multiple ascending dose (MAD) component. The goal of this study is to learn if GSM-779690T is safe and to assess the effects on levels of specific Aβ peptide isoforms in adults.

SAD: A total of 48 healthy volunteers are planned to be consented and enrolled to receive a single oral dose of GSM-779690T at increasing strengths or placebo in Cohorts 1 through 6.

MAD: A total of 48 healthy volunteers are planned to be consented and enrolled to receive multiple oral doses of GSM-779690T (doses will be informed by SAD data) in Cohorts 7 through 10. Cohort 10 will include healthy older-adults.

Participants who have signed an informed consent and meet screening eligibility requirements will be randomly assigned to receive a single oral dose of GSM-779690T or placebo with a 3:1 (active: placebo) ratio at each dose level. The decision to escalate between dose levels in the SAD and to proceed to the MAD will be based on Data Review Committee review of prior cohorts, safety, tolerability, and PK data. The study treatment, GSM-779690T, and all protocol assessments will be administered at the study site by trained study site personnel.

ELIGIBILITY:
Participants must meet all the following inclusion criteria to be eligible for enrollment:

1. Healthy, cognitively typical, and aged 20-45 years (inclusive).
2. Current Mini Mental State Examination (MMSE) score between 27 and 30 (inclusive) at screening.
3. Able to provide their own written informed consent.
4. Able to read, speak and understand English to ensure compliance with cognitive testing and study visit procedures.
5. Must be ambulatory and be willing to remain domiciled in the clinic for the required study procedures.
6. Contraception requirements:

   a. Women of childbearing potential (WOCBP) must agree to use a highly effective method of birth control (confirmed by the investigator) from enrollment, throughout the study duration, at 1 week after last dose of study treatment, and have a negative pregnancy test result at screening. Highly effective methods of birth control (those that can achieve a failure rate of less than 1% per year when used consistently and correctly) include: (i) Combined (oestrogen- and progestogen-containing) hormonal contraception associated with inhibition of ovulation: oral, intravaginal, or transdermal, (ii) Progestogen-only hormonal contraception associated with inhibition of ovulation: oral, injectable, or implantable, (iii) Intrauterine device, (iv) Intrauterine hormone-releasing system, (v) Bilateral tubal occlusion, (vi) Sexual abstinence, ie, refraining from heterosexual intercourse (vii) Vasectomised sexual partner (provided that partner is the sole sexual partner of the WOCBP study participants and that the vasectomized partner has received medical assessment of the surgical success).

   b. Women not of childbearing potential are defined as women who are either permanently sterilized (hysterectomy, bilateral oophorectomy, or bilateral salpingectomy) or who are postmenopausal. The following age-specific requirements apply: (i) Women < 50 years old will be considered postmenopausal if they have been amenorrhoeic for >12 months following cessation of exogenous hormonal treatment and FSH levels are in the postmenopausal range (>40 IU/L). Until FSH is documented to be within menopausal range, the patient should be treated as a WOCBP.

   (ii) Women > 50 years old will be considered postmenopausal if they have been amenorrhoeic for >12 months following cessation of all exogenous hormonal treatment.

   c. Males with childbearing partners must be willing to practice sexual abstinence or use double-barrier protection during study treatment and until 1 week after the last dose of study treatment.

   The same Inclusion Criteria as listed above for the phase 1A SAD study applies to the adult cohorts (aged 20-45 years, inclusive) in phase 1B MAD Study. The following additional inclusion criteria apply to the older-adult Cohort 10 only:

8. Healthy, cognitively typical, aged 60-75 years (inclusive).

9. Older participants (Cohort 10) must be living in the community (includes long-term assisted living facilities but excludes long-term care nursing facilities).

10. If applicable, older-adult participants (Cohort 10) diagnosed with chronic cardio- or metabolic diseases must have the condition well controlled (in the opinion of the investigator) to include a stable regimen for four (4) weeks prior to Dose Day 1. Some medications are permitted to treat common disorders, such as but not limited to hypertension, type II diabetes, dyslipidemia, and hypothyroidism.

11. Participants must have low likelihood of brain amyloid presence based on an amyloid probability score 2 (APS2) of < 47.5 calculated by PrecivityAD2™ test using the plasma sample collected at screening visit.

Participants meeting any of the following criteria must be excluded in the study:

1. History of any current or clinically significant gastrointestinal, renal, hepatic, bronchopulmonary, neurological, psychiatric, cardiovascular, endocrinological, ophthalmologic, hematological or allergic disease or metabolic disorder.

   Note: Older participants in Cohort 10 may be eligible if the chronic condition is well controlled per opinion of the clinical investigator.
2. Use of any concomitant medications is prohibited, other than prescribed birth control methods stable 4 weeks prior to screening.

   Note: Older participants in Cohort 10 who are taking stable dose regimen (4 weeks prior to Dose Day 1) may be eligible upon review and approval by the Medical Monitor.
3. A history of a psychiatric disorder such as schizophrenia, bipolar disorder or major depression according to the criteria of the most current version of the Diagnostic and Statistical Manual of Mental Disorders (DSM).
4. Any evidence of current suicidal ideation or any previous suicide attempt as evaluated by the Columbia-Suicide Severity Rating Scale (C-SSRS).
5. Diagnosis of a neurodegenerative disease or dementia, including but not limited to Alzheimer's disease (AD), Parkinson's disease and Huntington's disease.
6. A history of a seizure disorder.
7. Impaired hepatic function with any of the following lab abnormalities on screening:

   1. Alanine aminotransferase (ALT/SGPT) > 1.2X the upper limit of normal (ULN)
   2. Aspartate aminotransferase (AST/SGOT) values > 1.2X ULN
   3. Alkaline phosphatase (ALP) values > 1.2X ULN
   4. Total bilirubin > 1X ULN (excepting Gilbert's syndrome which is not an exclusion)
8. Renal function with an estimated glomerular filtration rate (eGFR) less than 90 mL/minute/1.73 m2 Note: less than 80 mL/minute/1.73 m2 in older participants enrolling in Cohort 10.
9. Presence of crystalluria in urinalysis at screening.
10. A clinically significantly abnormal 12-lead ECG result, including but not limited to: heart rate < 50 or > 100 beats per minute (bpm), QRS > 160 ms, QTcF > 450 ms in men & 460 ms in women, or any clinically significant arrhythmia including Mobitz type II second-degree atrioventricular (AV)(Hay block) block and bifascicular block.
11. A seated systolic blood pressure of < 100 or > 140 millimeters of mercury (mm Hg) or diastolic blood pressure of < 60 or > 90 mm Hg.

    1. Two readings should be taken approximately 1 minute apart and the average of the two will be applied.
    2. If the average is outside of the approved range, the procedure will be repeated following a brief rest.
12. Postural change at 3 min upon standing from seated position of:

    1. > 20 mm Hg systolic or > 10 mm Hg diastolic decrease in blood pressure
    2. > 30 bpm increase in heart rate
13. Cancer or malignant tumor within the past 3 years, except patients who underwent potentially curative therapy with no evidence of recurrence. Patients with stable untreated prostate cancer or skin cancers are not excluded.
14. Current acute or chronic Hepatitis A, B, C or HIV infection.
15. Alcohol abuse, alcohol dependence, or drug abuse in the past 5 years per most current version of the DSM.
16. Participation in another clinical trial with an investigational agent and have taken at least one dose of study medication, unless unblinded on placebo, within 3 months (12 weeks) or 5 drug half-lives (whichever is longer), prior to screening. (The end of a previous investigational trial is the date the last dose of an investigational agent was taken).
17. Previous treatment (within 1 year) with an investigational small molecule with anti-amyloid properties or passive immunization against Aβ or previous treatment with an active immunization against amyloid.
18. Positive result from a urine drug test at screening (screened for Amphetamines, Barbiturates, Cocaine metabolites, 3,4-Methylenedioxymethamphetamine (MDMA), Tricyclic Antidepressants (TCA), Phenylcyclohexyl Piperidine (PCP), Cotinine, Opiates, Benzodiazepines, Cannabinoids (THC), Methamphetamine, Methadone, Oxycodone (OXY)).
19. Not willing to abstain from consuming products containing caffeine (including chocolate), xanthine, citrus or alcohol from Day 1 through the end of the PK study.
20. SAD Cohorts 5, 6 and MAD Cohorts 9, 10: Contraindication to lumbar puncture (LP) This includes but is not limited to participants with a known allergy to the local anesthetics used in the LP, infection or inflammation of the skin or skin disease at or in proximity to the LP site; abnormal coagulation parameters, including platelet count, INR, PT and/or PTT, History of lumbar spine surgery or chronic low back pain for participants in the SAD Cohorts 5 and 6 and the MAD Cohorts 9 and 10.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-11-09 (Estimated); Primary Completion 2026-07-11 (Estimated); Study Completion 2026-07-11 (Estimated)

PRIMARY OUTCOMES:
Number and percentage of participants reporting treatment-emergent adverse events and serious adverse events after single and multiple oral doses of GSM-779690-T | From enrollment through study completion, approximately 7 days in groups 1, 2, 3, and 6; 14 days in groups 4 and 5; and 21 days in groups 7, 8, 9, and 10.
  Treatment emergent adverse events and serious adverse events will be summarized for each treatment group. The frequencies of treatment emergent adverse events and serious adverse events between the participants in each group will be compared.

OTHER OUTCOMES:
Pharmacokinetic parameter of area under the curve (AUC) calculation after single and multiple oral doses of GSM-779690-T | SAD Groups 1, 2, 3, 6 Days 0 to 7 post-dose (plasma); SAD Groups 4 and 5 Days 0 to 10 post-dose (plasma), Days 1 to 2 post-dose (CSF); MAD Groups 7, 8, 9 and 10 Days 0 to 16 post-dose (plasma), Days 14 to 15 post-dose (CSF).
• Pharmacokinetic Parameter of maximum plasma concentration (cmax) calculation after single and multiple oral doses of GSM-779690-T | SAD Groups 1, 2, 3, 6 Days 0 to 7 post-dose (plasma); SAD Groups 4 and 5 Days 0 to 10 post-dose (plasma), Days 1 to 2 post-dose (CSF); MAD Groups 7, 8, 9 and 10 Days 0 to 16 post-dose (plasma), Days 14 to 15 post-dose (CSF).
Pharmacokinetic Parameter of time to maximum plasma concentration (tmax) calculation after single and multiple oral doses of GSM-779690-T | SAD Groups 1, 2, 3, 6 Days 0 to 7 post-dose (plasma); SAD Groups 4 and 5 Days 0 to 10 post-dose (plasma), Days 1 to 2 post-dose (CSF); MAD Groups 7, 8, 9 and 10 Days 0 to 16 post-dose (plasma), Days 14 to 15 post-dose (CSF).

CONTACTS AND LOCATIONS:
Overall Officials: Doug Galasko, MD, Principal Investigator — University of California, San Diego
Locations (1):
- Worldwide Clinical Trials, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: No